CLINICAL TRIAL: NCT01132105
Title: Vestibular Evoked Myogenic Potential: A New Device Propose
Status: Completed | Type: Observational
Sponsor: Universidade Estadual de Ciências da Saúde de Alagoas (Other)
Collaborators: Aline Carabl de Oliveira (Unknown); José Fernando Colafêmina (Unknown)
Other Study IDs: UNCISAL-PM-001
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Evoked Potentials, Motor, Vestibular

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Normal subjects: Adults normal hearing and vestibular function subjects
  Interventions: Device: Vestibular myogenic evoked potential analyzer

INTERVENTIONS:
Device: Vestibular myogenic evoked potential analyzer

SUMMARY:
The bioelectrical responses of muscle, evoked by sound, obtained with a device considered the gold standard (widely used in clinics and hospitals) are similar to those obtained with a new device developed

ELIGIBILITY:
Inclusion Criteria:

* hearing thresholds equal to or less than 20 dB HL with differences between the ears, by frequency, equal to or less than 10 dB.

Exclusion Criteria:

* Occupational noise exposure
* Ear surgeries
* More than three ear infections in the current year
* Use of ototoxic medication
* Tinnitus, vertigo, dizziness or other vestibular-cochlear diseases
* Systemic diseases that may contribute to cochlear-vestibular pathologies, such as hypertension and dyslipidemia
* Hormonal diseases

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults, Normal Hearing, Normal Vestibular fuction,
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Menezes, PhD, Principal Investigator — Universidade Estadual de Ciências da Saúde de Alagoas
Locations (1):
- Universidade Estadual de Ciências da Saúde de Alagoas - UNCISAL, Maceió, Alagoas, Brazil